CLINICAL TRIAL: NCT03882333
Title: Effects of Acute Exercise on Pain and Human Movement - a Randomised Controlled Study in Patients With Chronic Pain and Healthy Controls
Brief Title: Effects of Acute Exercise on Pain and Human Movement
Acronym: eMOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna University (Other)
Collaborators: Dalarna County Council, Sweden (Other); Swedish Council for Working Life and Social Research (Other); Karolinska Institutet (Other); Swedish Armed Forces (Unknown)
Responsible Party: Principal Investigator, Bjorn Ang, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dalarna University 2017-00177
Record Dates: First submitted 2018-12-12; First posted 2019-03-20 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Chronic Musculoskeletal Disease; Chronic Pain, Widespread
Keywords: Chronic musculoskeletal pain; Acute exercise; Movement control; Muscle activity
MeSH Terms: conditions — Chronic Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A randomised controlled study in patients with chronic pain and healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute exercise (Experimental): Acute exercise (bicycle at stationary cycle).
  Interventions: Other: Acute exercise
- Rest (No Intervention): Rest (lying down or sitting in a chair) for 30 minutes, i.e. same time duration as in experimental arm.

INTERVENTIONS:
Other: Acute exercise — 30 min acute exercise (bicycle at stationary cycle)
  Arms: Acute exercise

SUMMARY:
The aim of this research project is to evaluate the effect of an acute exercise intervention on pain intensity and movement control. It also aims to investigate potential differences in movement con-trol between patients with chronic musculoskeletal pain compared to healthy controls.

DETAILED DESCRIPTION:
The aim of this research project is to evaluate the effect of an acute exercise intervention on pain intensity and movement control. It also aims to investigate potential differences in movement control between patients with chronic musculoskeletal pain compared to healthy controls. All tests will be conducted at Dalarna University.

After the initial baseline tests, participants will be randomised to either acute exercise intervention group or to a control group not performing any intervention groups (both patients and controls will be randomised to intervention or control). If randomised to the control group, participants rests corresponding to the time it takes to perform the intervention (30 min), and then preform the post-intervention tests similar as the intervention group.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for participants with chronic pain:

* Men and women, age 18-67 years,
* good ability to understand written and verbal information and instruction given in Swedish,
* chronic (>3 months) musculoskeletal pain or chronic widespread pain.

Inclusion criteria for healthy controls:

* Men and women, age 18-67 years,
* good ability to understand written and verbal information and instruction given in Swedish.

Exclusion Criteria:

For participants with chronic pain

* chronic pain caused by malignancies or systemic diseases, other physical conditions that affects functional abilities and implies use of walking aid in-door,
* pregnancy after week 12, childbirth within the last 3 months or
* spinal surgery.

For healthy controls:

* chronic (>3 months) or acute pain of any cause,
* other physical conditions that affects functional abilities, and implies use of walking aids in-door,
* pregnancy after week 12, childbirth in the last 3 months or
* spinal surgery.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Kinematic measures of human movement during functional gait sequences | 30 minutes (before and after the acute exercise intervention)
  Objective measures of movement control using sophisticated wearable sensors (accelerometer-based APDM-sensors applied at participants wrists, ankles, chest and head) during walking in 1) self-selected normal gait speed, 2) a brisk gait speed, 3) self-selected normal gait speed with a concurrent cognitive task (1-back test: participants listens to a recording of a voice that presents random series of digits between 1 to 9 with two seconds apart. The participants will be instructed to respond as quickly and accurately as possible, repeating the digit before the last one in the sequence.). Lumbar trunk rotations (degrees) will specifically be evaluated while many other kinematic variables (walking speed, step length, step width etc) will be analyzed with factor analyz-es to reduce data variables to relevant data domains, such as gait stability. Data will be aggregated as means and variances.
Muscle activity | 30 minutes (before and after the acute exercise intervention)
  Evaluation of back muscle activity using electromyographics (EMG) during walking as in outcome 1, i.e. in 1) self-selected normal gait speed, 2) a brisk gait speed, 3) self-selected normal gait speed with a concurrent cognitive task (1-back test). Participants will be instrumented with surface-EMG (Delsys Incorporated, Massachusetts) electrodes applied bilateral at participants back and neck muscles. Back and neck spatial and temporal muscle activity (EMG amplitudes) representing repeated gait cycles will be aggregated to one cycle; factor analyzes may be applied to reduce data variables to relevant data domains. Data will be presented as means and variances.

SECONDARY OUTCOMES:
Self-rated pain using the Visual Analogue Scale (VAS scale). | 30 minutes (before and after the acute exercise intervention)
  Self-rated pain will be measured using a horizontal 10-cm line "Visual Analogue Scale" (VAS) with the statement 'no pain at all' at the extreme left-hand end, and 'the worst possible pain' or 'unbearable' at the right-hand extreme.

CONTACTS AND LOCATIONS:
Overall Officials: Björn BA Äng, Assoc. Prof., Principal Investigator — Dalarna University
Locations (1):
- Dalarna University (LIVI lab), Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boecker H, Sprenger T, Spilker ME, Henriksen G, Koppenhoefer M, Wagner KJ, Valet M, Berthele A, Tolle TR. The runner's high: opioidergic mechanisms in the human brain. Cereb Cortex. 2008 Nov;18(11):2523-31. doi: 10.1093/cercor/bhn013. Epub 2008 Feb 21. PMID 18296435
- [Background] Brumagne S, Janssens L, Knapen S, Claeys K, Suuden-Johanson E. Persons with recurrent low back pain exhibit a rigid postural control strategy. Eur Spine J. 2008 Sep;17(9):1177-84. doi: 10.1007/s00586-008-0709-7. Epub 2008 Jul 2. PMID 18594876
- [Background] van den Hoorn W, Bruijn SM, Meijer OG, Hodges PW, van Dieen JH. Mechanical coupling between transverse plane pelvis and thorax rotations during gait is higher in people with low back pain. J Biomech. 2012 Jan 10;45(2):342-7. doi: 10.1016/j.jbiomech.2011.10.024. Epub 2011 Nov 10. PMID 22078275
- [Background] Seay JF, Van Emmerik RE, Hamill J. Influence of low back pain status on pelvis-trunk coordination during walking and running. Spine (Phila Pa 1976). 2011 Jul 15;36(16):E1070-9. doi: 10.1097/BRS.0b013e3182015f7c. PMID 21304421
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Darnall BD, Sturgeon JA, Cook KF, Taub CJ, Roy A, Burns JW, Sullivan M, Mackey SC. Development and Validation of a Daily Pain Catastrophizing Scale. J Pain. 2017 Sep;18(9):1139-1149. doi: 10.1016/j.jpain.2017.05.003. Epub 2017 May 19. PMID 28528981
- [Background] Bergstrom G, Jensen IB, Bodin L, Linton SJ, Nygren AL, Carlsson SG. Reliability and factor structure of the Multidimensional Pain Inventory--Swedish Language Version (MPI-S). Pain. 1998 Mar;75(1):101-110. doi: 10.1016/S0304-3959(97)00210-8. PMID 9539679
- [Background] Tseli E, Boersma K, Stalnacke BM, Enthoven P, Gerdle B, Ang BO, Grooten WJA. Prognostic Factors for Physical Functioning After Multidisciplinary Rehabilitation in Patients With Chronic Musculoskeletal Pain: A Systematic Review and Meta-Analysis. Clin J Pain. 2019 Feb;35(2):148-173. doi: 10.1097/AJP.0000000000000669. PMID 30371517
- [Background] Molander P, Dong HJ, Ang B, Enthoven P, Gerdle B. The role of pain in chronic pain patients' perception of health-related quality of life: a cross-sectional SQRP study of 40,000 patients. Scand J Pain. 2018 Jul 26;18(3):417-429. doi: 10.1515/sjpain-2018-0003. PMID 29794267
- [Derived] Westergren J, Sjoberg V, Vixner L, Nyberg RG, Moulaee Conradsson D, Monnier A, LoMartire R, Enthoven P, Ang BO. Acute exercise as active inference in chronic musculoskeletal pain, effects on gait kinematics and muscular activity in patients and healthy participants: a study protocol for a randomised controlled laboratory trial. BMJ Open. 2023 May 31;13(5):e069747. doi: 10.1136/bmjopen-2022-069747. PMID 37258077